CLINICAL TRIAL: NCT02786511
Title: Longterm Follow-up of Subjects Treated With bb2121
Status: Completed | Type: Observational
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Other Study IDs: LTF-305
Record Dates: First submitted 2016-05-26; First posted 2016-06-01 (Estimated); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Safety

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subjects with multiple myeloma: Subjects treated with ex vivo gene therapy in a bluebird bio sponsored trial who agree to participate in this study.
  Interventions: Drug: Safety and efficacy assessments

INTERVENTIONS:
Drug: Safety and efficacy assessments — Vector copy number (VCN) measurement, safety evaluations, disease-specific assessments, and assessments to monitor for long-term implications of autologous transplant

SUMMARY:
This is a multi-center, non-randomized, open label, longterm safety and efficacy follow-up study for subjects who have been treated with bb2121 in the Phase 1 clinical parent study, that evaluated the safety and efficacy of bb2121 in subjects with relapsed or refractory B cell maturation antigen (BCMA)-expressing multiple myeloma.

bb2121 is defined as autologous T lymphocytes (T cells) transduced ex vivo with anti-BCMA02 CAR lentiviral vector encoding the chimeric antigen receptor (CAR) targeted to human BCMA suspended in cryopreservative solution. bb2121 is administered in subjects 1 time (or retreated if retreatment criteria are met) in parent clinical study. No investigational treatment will be administered in this study.

After completing the parent study, eligible subjects will be followed for up to 15 years after their last bb2121 infusion in the parent study.

DETAILED DESCRIPTION:
The LTF-305 study has completed enrollment and is scheduled to be closed. All patients participating in this study have discontinued from follow-up or have been transferred into the GC-LTFU-001 study for further observation (similar to time frames established in the LTF-305).

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent for this study by subjects
* Were administered bb2121 in the parent clinical study
* Able to comply with the study requirements

Exclusion Criteria:

* Subject has disease progression AND subject has undetectable VCN (<0.0003 vector copies per diploid genome) in peripheral blood cells for 2 consecutive measurements at least 1 month apart, at least 12 months after drug product infusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with multiple myeloma who were administered bb2121 in Study CRB-401
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-04-28 (Actual); Primary Completion 2019-10-11 (Actual); Study Completion 2019-10-11 (Actual)

PRIMARY OUTCOMES:
Overall survival | 15 years post-drug product infusion
Monitoring for all Adverse Events, including Serious Adverse Events, related to the drug product | 15 years post-drug product infusion
Monitoring for all Serious Adverse Events including any new malignancy or new diagnosis of a neurologic, rheumatologic, or hematologic disorder that is clinically significant | 5 years post-drug product infusion
Monitoring for Multiple Myeloma-specific response according to the International Myeloma Working Group (IMWG) Uniform Response Criteria for Multiple Myeloma | 5-15 years post-drug product infusion
  Subjects without disease progression will be evaluated for at least 5 years post-drug product infusion if VCN is undetectable, and up to 15 years post-drug product infusion if VCN remains detectable.
Progression Free Survival | 5-15 years post-drug product infusion
  Subjects without disease progression will be evaluated for at least 5 years post-drug product infusion if VCN is undetectable, and up to 15 years post-drug product infusion if VCN remains detectable.
Monitoring for Vector Copy Number (VCN) | 5-15 years post-drug product infusion
  Subjects without disease progression will be evaluated for at least 5 years post-drug product infusion if VCN is undetectable, and up to 15 years post-drug product infusion if VCN remains detectable.

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Hege, Study Director — Celgene Corporation
Locations (9):
- United States (9):
  - Stanford Cancer Center, Palo Alto, California
  - National Cancer Institute, Bethesda, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Mount Sinai Medical Center, New York, New York
  - Sarah Cannon Research Institute, Nashville, Tennessee